CLINICAL TRIAL: NCT03496675
Title: Music Interventions for Dementia and Depression in Elderly Care: International Cluster-randomised Controlled Trial
Brief Title: Music Interventions for Dementia and Depression in Elderly Care
Acronym: MIDDEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NORCE Norwegian Research Centre AS (Other)
Collaborators: University of Melbourne (Other); University of Oldenburg (Other); University Medical Center Groningen (Other); Ankara Haci Bayram Veli University (Unknown); University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: MIDDEL
Record Dates: First submitted 2018-03-06; First posted 2018-04-12 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Dementia; Depression
MeSH Terms: conditions — Dementia; Depression | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinding of assessors will be ensured by using assessors who do not participate in the daily care of each unit. Assessors will also remind participants not to reveal the unit's allocation to them. At the time of the last assessment, success of blinding will be verified by asking assessors whether they inadvertently discovered the unit's allocation. Intervention providers and study participants (PLWD and staff) cannot be blinded due to the nature of the interventions. However, efforts will be made to ensure that no differential expectations are created and equipoise is maintained (e.g., by careful wording of the patient information and consent form).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Standard care (Other): Participants receive standard care as locally available. The components of standard care are recorded.
  Interventions: Other: Standard care
- Group Music Therapy (GMT) (Experimental): GMT is provided twice weekly for the first three months, followed by weekly sessions for the next three months, with possible extension after that period as desired and feasible. Sessions are 45 minutes each.
  In line with usual practice, and as appropriate in local contexts, residents of a unit allocated to GMT may be divided into smaller groups (e.g. around 5 participants).
  Interventions: Behavioral: Group Music Therapy; Other: Standard care
- Recreational Choir Singing (RCS) (Experimental): RCS is provided twice weekly for the first three months, followed by weekly sessions for the next three months, with possible extension after that period as desired and feasible. Sessions are 45 minutes each.
  RCS may be conducted in larger groups (e.g. with all residents of the unit in one group).
  Interventions: Behavioral: Recreational Choir Singing; Other: Standard care
- GMT + RCS (Experimental): Group Music Therapy and Recreational Choir Singing are both provided twice weekly for the first three months, followed by weekly sessions for the next three months, with possible extension after that period as desired and feasible. Sessions are 45 minutes each.
  Interventions: Behavioral: Group Music Therapy; Behavioral: Recreational Choir Singing; Other: Standard care

INTERVENTIONS:
Behavioral: Group Music Therapy — The core intention of GMT is to meet the psychosocial needs of each person living with dementia, which in turn is thought to reduce depressive symptoms and anxiety and to stimulate overall social and emotional wellbeing. It includes active, reciprocal music making with the use of singing and musical instruments. GMT is provided by a trained music therapist, highly skilled as a musician, and registered with the appropriate professional association in his or her country.
  Arms: GMT + RCS; Group Music Therapy (GMT)
Behavioral: Recreational Choir Singing — RCS is intended to foster connectedness in a group, wellbeing, and enjoyment of music making in a group. It includes singing familiar songs and providing a familiar musical environment for participants. RCS is provided by a musician with choir leading skills.
  Arms: GMT + RCS; Recreational Choir Singing (RCS)
Other: Standard care — May include pharmacological and non-pharmacological interventions as locally available

SUMMARY:
This study evaluates the effectiveness of two music-based approaches - group music therapy and recreational choir singing - for reducing depression symptoms in people living with dementia. It also examines mechanisms and heterogeneity of treatment effects.

DETAILED DESCRIPTION:
Dementia and depression are highly prevalent and comorbid conditions in older adults and are associated with individual distress, substantial carer burden, and high societal costs.

Music interventions represent a highly promising type of non-pharmacological interventions for both dementia and depression in older adults. They are widely used, but have yet to be rigorously tested in large trials.

The MIDDEL trial is the largest trial of music interventions to date, and the first to compare different music-based interventions - group music therapy (GMT), and recreational choir singing (RCS) - alone and in combination across countries.

MIDDEL is designed as a large, pragmatic, international cluster-randomised controlled trial with a 2x2 factorial design that will compare the effects of GMT, RCS, both, or neither, for care home residents aged 65 years or older with dementia and depressive symptoms.

Study sites will be located in Australia and in five European countries, and a total of 100 care home units will be randomised to one of the four study conditions.

ELIGIBILITY:
Inclusion Criteria:

* resident (full-time, 24h/day) at a participating care home;
* dementia as indicated by a Clinical Dementia Rating score of 0.5 or more and a Mini-Mental State Examination (MMSE) score of 26 or less;
* at least mild depressive symptoms, as indicated by a Montgomery-Åsberg Depression Rating Scale (MADRS) score of at least 8;
* a clinical diagnosis of dementia according to ICD-10 research criteria;
* have given written informed consent (may be assent by proxy for those unable to provide consent themselves).

Exclusion Criteria:

* diagnosis of schizophrenia or Parkinson's disease;
* severe hearing-impairment;
* in short-term care;
* unable to tolerate sitting in a chair for the duration of the sessions.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1021 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) | 6 months
  10-item scale where each item is rated from 0 to 6 ('no abnormality' to 'severe'), yielding a total sum score between 0 and 60, with higher values indicating more severe symptom levels.

SECONDARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) | up to 24 months
  10-item scale where each item is rated from 0 to 6 ('no abnormality' to 'severe'), yielding a total sum score between 0 and 60, with higher values indicating more severe symptom levels.
Clinical Dementia Rating (CDR) | 12 months
  Semi-structured interview with the person living with dementia and an appropriate caregiver/relative; rates impairment across 6 cognitive categories (memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care). The CDR score can range from 0 (normal) to 3 (severe dementia); not used at all sites.
Neuropsychiatric Inventory - Questionnaire (NPI-Q): severity | 12 months
  Includes 12 domains where if a symptom is present, its severity (from 1 = mild to 3 = severe) is assessed by a caregiver familiar with the participant's behaviour. Higher scores (sums of all items, range 0 to 36) represent higher severity.
Neuropsychiatric Inventory - Questionnaire (NPI-Q): distress | 12 months
  Includes 12 domains where if a symptom is present, the associated distress on caregivers (from 0 = not distressing at all to 5 = extreme or very severe) is assessed by a caregiver familiar with the participant's behaviour. Higher scores (sums of all items, range 0 to 60) represent higher severity.
EuroQol (EQ-5D) | 12 months
  Standardized, non-disease-specific instrument for evaluating health-related quality of life, defining health in five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Response categories range from "no problems" to "extreme problems". Scores are derived using a weighted scoring method and can range from 0 = worst possible to 1 = best possible quality of life.
Quality of Life in Alzheimer´s Dementia (QOL-AD) | 12 months
  13-item scale with self-rating and proxy version. Each item ranges from 1 (poor) to 4 (excellent), yielding a total sum score of 13 to 52.
All-cause mortality (time to death) | up 24 months
  Data on participant deaths will be collected from care staff on a monthly basis.
Any increase in medication use (binary, yes/no) | 12 months
  Data on type (ATC Codes N065, N06) of medication used and any increase or decrease over time will be collected from care staff using the 'medication profile' section of a tailored version of the Client Socio-Demographic and Service Receipt Inventory (CSSRI), or from available databases.
Costs | 12 months
  Total and component costs of the interventions are assessed from a societal perspective, including the cost of the intervention as well as statutory health and social care services used, using a tailored version of the Client Socio-Demographic and Service Receipt Inventory (CSSRI). Total cost per participant will be calculated in Euros.
Any adverse event [Safety] | 12 months
  All types of adverse events and serious adverse events (e.g. unexpected worsening of symptoms), whether related or unrelated to the interventions, are reported.
Professional Care Team Burden Scale | 12 months
  10-item scale to obtain ratings of burden from formal care teams working in care homes. Items are scored on a 5-point scale from 0 (strongly disagree) to 4 (strongly agree), yielding a total sum score from 0 to 40, with higher scores indicating higher burden.
Days on sick leave of care staff | 12 months
  (as recorded monthly by the employer)

CONTACTS AND LOCATIONS:
Overall Officials: Vigdis Sveinsdottir, PhD, Principal Investigator — GAMUT, NORCE Norwegian Research Centre, Bergen, Norway
Locations (6):
- The University of Melbourne, Melbourne, Victoria, Australia
- Carl von Ossietzky University Oldenburg, Oldenburg, Germany
- University Medical Centre Groningen, Groningen, Netherlands
- NORCE Norwegian Research Centre, Bergen, Vestland, Norway
- Ankara Hacı Bayram Veli University, Ankara, Turkey (Türkiye)
- University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified datasets (participant codes and outcome scores) generated during and/or analysed during the current study will be stored in a publically available repository (NSD - Norwegian Centre for Research Data, http://www.nsd.uib.no/nsd/english/index.html).
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will become available upon publication of the primary outcome.
Access Criteria: De-identified IPD will be publicly available at the Norwegian Centre for Research Data (http://www.nsd.uib.no/nsd/english/index.html).

REFERENCES:
- [Background] Janus, S. I. M., Vink, A. C., Ridder, H. M., Geretsegger, M., Stige, B., Gold, C., & Zuidema, S. U. (2020). Developing consensus description of group music therapy characteristics for persons with dementia. Nordic Journal of Music Therapy, 1-17.
- [Background] Baker FA, Tamplin J, Clark IN, Lee YC, Geretsegger M, Gold C. Treatment Fidelity in a Music Therapy Multi-site Cluster Randomized Controlled Trial for People Living With Dementia: The MIDDEL Project Intervention Fidelity Protocol. J Music Ther. 2019 May 10;56(2):125-148. doi: 10.1093/jmt/thy023. PMID 30721998
- [Background] Baker FA, Lee YC, Sousa TV, Stretton-Smith PA, Tamplin J, Sveinsdottir V, Geretsegger M, Wake JD, Assmus J, Gold C. Clinical effectiveness of music interventions for dementia and depression in elderly care (MIDDEL): Australian cohort of an international pragmatic cluster-randomised controlled trial. Lancet Healthy Longev. 2022 Mar;3(3):e153-e165. doi: 10.1016/S2666-7568(22)00027-7. PMID 36098290
- [Background] Baker FA, Stretton-Smith PA, Sousa TV, Clark I, Cotton A, Gold C, Lee YC. Resource assessment in trials undertaken in residential care homes: Experiences from the Australian MIDDEL cluster randomised controlled trial research team. Contemp Clin Trials Commun. 2020 Nov 25;20:100675. doi: 10.1016/j.conctc.2020.100675. eCollection 2020 Dec. PMID 33305065
- [Background] Gold C, Eickholt J, Assmus J, Stige B, Wake JD, Baker FA, Tamplin J, Clark I, Lee YC, Jacobsen SL, Ridder HMO, Kreutz G, Muthesius D, Wosch T, Ceccato E, Raglio A, Ruggeri M, Vink A, Zuidema S, Odell-Miller H, Orrell M, Schneider J, Kubiak C, Romeo R, Geretsegger M. Music Interventions for Dementia and Depression in ELderly care (MIDDEL): protocol and statistical analysis plan for a multinational cluster-randomised trial. BMJ Open. 2019 Mar 30;9(3):e023436. doi: 10.1136/bmjopen-2018-023436. PMID 30928926
- [Background] Lee YC, Sousa TV, Stretton-Smith PA, Gold C, Geretsegger M, Baker FA. Demographic and clinical profile of residents living with dementia and depressive symptoms in Australian private residential aged care: Data from the Music Interventions for Dementia and Depression in ELderly care (MIDDEL) cluster-randomised controlled trial. Australas J Ageing. 2022 Dec;41(4):e387-e396. doi: 10.1111/ajag.13104. Epub 2022 Jul 8. PMID 35801957
- [Background] Rasing NL, Janus SIM, Kreutz G, Sveinsdottir V, Gold C, Nater UM, Zuidema SU. The Impact of Music on Stress Biomarkers: Protocol of a Substudy of the Cluster-Randomized Controlled Trial Music Interventions for Dementia and Depression in ELderly Care (MIDDEL). Brain Sci. 2022 Apr 8;12(4):485. doi: 10.3390/brainsci12040485. PMID 35448016
- [Derived] Schneider J, Ablewhite J, Bloska J, Orrell M, Odell-Miller H, Assmus J, Gold C, Sveinsdottir V. Impact of Music Interventions on Depression in Care Home Residents with Dementia: UK Results from Music Interventions for Depression and Dementia in Elderly Care RCT. Geriatrics (Basel). 2025 Dec 15;10(6):166. doi: 10.3390/geriatrics10060166. PMID 41440736
- [Derived] Sveinsdottir V, Assmus J, Schneider J, Baker FA, Ucaner B, Kreutz G, Geretsegger M, Rasing N, Bloska J, Stretton-Smith PA, Lee YC, Wake JD, Odell-Miller H, Tamplin J, Vink AC, Ablewhite J, Neuser J, Frischen U, Timmer A, Wosch T, Janus S, Gold C. Clinical effectiveness of music interventions for dementia and depression in older people (MIDDEL): a multinational, cluster-randomised controlled trial. Lancet Healthy Longev. 2025 Dec;6(12):100783. doi: 10.1016/j.lanhl.2025.100783. Epub 2025 Dec 8. PMID 41380710
- [Derived] Rasing NL, Janus SIM, Vink AC, Frischen UAS, Neuser J, Wake JD, Skoluda N, Sveinsdottir V, Geretsegger M, Langeland E, Kreutz G, Gold C, Nater UM, Zuidema SU. The short-term impact of music interventions on stress: Results of a multinational cluster-randomized trial using salivary cortisol and alpha-amylase assessments in care home residents with dementia. Psychoneuroendocrinology. 2025 Dec;182:107640. doi: 10.1016/j.psyneuen.2025.107640. Epub 2025 Oct 2. PMID 41072366
- [Derived] Rasing NL, Vink AC, Bloska J, Nevruz H, Bakirci T, Saltik Y, Ucaner B, Dugstad Wake J, Sveinsdottir V, Geretsegger M, Gold C, Frischen U, Neuser J, Kreutz G, Zuidema SU, Janus SIM. Video Analysis of Group Music Therapy for Dementia: Intervention Delivery and Treatment Fidelity. J Music Ther. 2025 Jan 10;62(1):thaf007. doi: 10.1093/jmt/thaf007. PMID 40616479
- See also: Project website — http://middel-project.eu
- Available data/document: Individual Participant Data Set — https://osf.io/tpdhu/